CLINICAL TRIAL: NCT06248320
Title: Effect of Perioperative Sigh Ventilation on Postoperative Hypoxemia and Pulmonary Complications After On-pump Cardiac Surgery: A Randomized Controlled Trial
Brief Title: Sigh Ventilation on Postoperative Hypoxemia in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Fengmei Guo, Director of Intensive Care Unit, Principal Investigator, Clinical Professor, Zhongda Hospital, Southeast University, China, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIGHVENT
Record Dates: First submitted 2024-01-30; First posted 2024-02-08 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Hypoxemia; Postoperative Complications; Cardiac Disease; Acute Lung Injury
Keywords: Mechanical ventilation; Cardiac Surgery; Hypoxemia; Pulmonary Complications
MeSH Terms: conditions — Hypoxia; Postoperative Complications; Heart Diseases; Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sigh ventilation (Experimental): * Sigh breaths consisting of increasing positive end-expiratory pressure (PEEP) that produces a plateau pressure of 35 cmH2O (or 40 cmH2O in patients with BMIs > 35). The sigh breaths will be delivered once every 6 minutes, as part of usual invasive mechanical ventilation, from intubation to extubation.
  * No sigh ventilation during thoracotomy
  * Lung protective ventilation from intubation to extubation, consisted of low tidal volume (6-8ml/kg/pbw) and positive end-expiratory pressure setting according to ARDS low PEEP-FiO2 table
  Interventions: Procedure: Sigh ventilation
- Conventional ventilation (No Intervention): - Lung protective ventilation from intubation to extubation, consisted of low tidal volume (6-8ml/kg/pbw) and positive end-expiratory pressure setting according to ARDS low PEEP-FiO2 table

INTERVENTIONS:
Procedure: Sigh ventilation — Sigh breaths were delivered from intubation to extubation. Intervention primarily conducted in the following three stages: 1. From intubation to surgical opening of the chest cavity; 2. From the surgical closure of the chest cavity close and continue unit the operating room exiting; 3. From Intensive Care Unit (ICU) arrival to Spontaneous breathing trial (SBT) start.
  Arms: Sigh ventilation

SUMMARY:
Postoperative pulmonary complications (PPCs) remain a frequent event after pump-on cardiac surgery and are mostly characterized by postoperative hypoxemia.These complications are significant contributors to prolonged intensive care unit admissions and an escalation in in-hospital mortality rates.

The dual impact of general anesthesia with invasive mechanical ventilation results in ventilator-induced lung injury, while cardiac surgery introduces additional pulmonary insults. These include systemic inflammatory responses initiated by cardiopulmonary bypass and ischemic lung damage consequent to aortic cross-clamping. Contributing factors such as blood transfusions and postoperative pain further exacerbate the incidence of PPCs by increasing the permeability of the alveolar-capillary barrier and disrupting mucociliary functions, often culminating in pulmonary atelectasis.

Protective ventilation strategies, inspired by acute respiratory distress syndrome (ARDS) management protocols, involve the utilization of low tidal volumes (6-8mL/kg predicted body weight). However, the uniform application of low tidal volumes, especially when combined with the multifactorial pulmonary insults inherent to cardiac surgery, can precipitate surfactant dysfunction and induce atelectasis.

The role of pulmonary surfactant in maintaining alveolar stability is critical, necessitating continuous synthesis to sustain low surface tension and prevent alveolar collapse. The most potent stimulus for surfactant secretion is identified as the mechanical stretch of type II pneumocytes, typically induced by larger tidal volumes.

This background sets the foundation for a research study aimed at assessing the safety and efficacy of incorporating sighs into perioperative protective ventilation. This approach is hypothesized to mitigate postoperative hypoxemia and reduce the incidence of PPCs in patients undergoing scheduled on-pump cardiac surgery.

DETAILED DESCRIPTION:
The purpose of this single center, parallel group, randomized controlled study is to evaluate the effect of a perioperative sigh ventilation strategy on postoperative outcomes during the first 7 days following cardiac surgery. The study will include 192 adult patients undergoing scheduled on-pump cardiac surgery. The sigh ventilation approach will combine sigh ventilation and lung protective ventilation (6-8 ml/kg/pbw) from intubation to extubation. It will be compared to a conventional approach without sigh ventilation, with lung protective ventilation and positive end-expiratory pressure (PEEP) setting same as the intervention arm. The primary endpoint is the Spo2/Fio2 ratio during the initial post extubation hour. The secondary endpoints are postoperative pulmonary complications and hospital length of stay .

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery with general anesthesia
* Conventional cardiopulmonary bypass and aortic cross clamp
* Providing written informed consent by the patient himself/herself or the next of kin

Exclusion Criteria:

* Emergent surgery including aortic dissection, cardiac rupture and active endocarditis surgery
* Left ventricular assist device implantation
* Patients anticipated to require intraoperative support with Extracorporeal Membrane Oxygenation (ECMO) or Intra-Aortic Balloon Pump (IABP)
* Chronic pulmonary disease requiring long-term home oxygen therapy
* Receiving invasive mechanical ventilation within 7 days prior to surgery
* Preoperative shock
* Obstructive Sleep Apnea Syndrome (OSAS) requiring intermittent non-invasive ventilatort support
* Preoperative left ventricular ejection fraction<40%
* Pulmonary arterial systolic pressure>50 mmHg
* Redo surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
Time-weighted average pulse oximetry (SpO2/FiO2) | 1 hour after endotracheal extubation
  Calculated the SpO2/FiO2 ratio every 15min during the initial postextubation hour, then averaged the SpO2/FiO2 ratios weighted by measurement interval. The comparison between arms was made through T-test.

SECONDARY OUTCOMES:
Proportion of respiratory failure | first 7 days postextubation
  Mild respiratory failure: SpO2 < 90% or PaO2 < 60 mmHg after breathing ambient air for 10 min (excluding hypoventilation) and corrected with an oxygen supply of 1-3 L/min with a nasal cannula; Moderate respiratory failure: SpO2 < 90% or PaO2 < 60 mmHg despite a 3 L/min oxygen supply with a nasal cannula (excluding hypoventilation) and corrected with an oxygen supply from 4 to 10 L/ min with a face mask; Severe respiratory failure: SpO2 < 90% or PaO2 < 60 mmHg despite a 10 L/min oxygen supply with a face mask (excluding hypoventilation) and corrected with an oxygen supply > 10 L/min with a high-flow face mask or with non-invasive ventilation or with high-flow nasal oxygen therapy or with invasive mechanical ventilation. Using the worst score in the first 7 days postextubation for main analysis.
  Tested between arms through ordinal logistic regression.
Severity of postoperative pulmonary complications | first 7 days after surgery
  Score of pulmonary complications adapted from previous publications, with 5 degrees, where the higher one means death before hospital discharge, degree (4) means the need of mechanical ventilation for more than 48 hours after surgery or after reintubation, degree (3) means pneumonia or intense noninvasive ventilation need, degree (2) means hypoxemia and abnormal lung findings, degree 1 means simple atelectasis and degree (0) means no complication. Using the worst score in the first 7 days after surgery for main analysis.
  Tested between arms through ordinal logistic regression.
Invasive mechanical ventilation (IMV) days | first 7 days after surgery
  Durations of invasive mechanical ventilation.
Reintubation rate | first 7 days after surgery
  Occurrence of endotracheal reintubation.
Proportion of receiving non-invasive ventilation (NIV) or High-flow nasal cannula (HFNC) support | first 7 days after surgery
  Tested through the Fisher exact test or chi-square test.
No ventilatory-support days | first 7 days after surgery
  Days alive and not receive IMV, HFNC and non-invasive ventilatory support.
In-hospital mortality | From the day of surgery up to Hospital discharge or death, maximum censoring at day 28 after surgery
  Deaths occurred during hospital stay
Length of ICU stay | From the day of surgery up to ICU discharge, maximum censoring at day 28 after surgery
  Days since surgery until ICU discharge
Length of hospital stay | From the day of surgery up to Hospital discharge, maximum censoring at day 28 after surgery
  Days since surgery until Hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Fengmei Guo, PhD, MD, Study Chair — Nanjing Zhongda Hospital, Southeast University
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Z, Cheng Q, Huang S, Sun J, Xu J, Xie J, Cao H, Guo F. Effect of perioperative sigh ventilation on postoperative hypoxemia and pulmonary complications after on-pump cardiac surgery (E-SIGHT): study protocol for a randomized controlled trial. Trials. 2024 Sep 4;25(1):585. doi: 10.1186/s13063-024-08416-y. PMID 39232795